CLINICAL TRIAL: NCT06788782
Title: Retrospective Analysis of Candida-associated Osteoarticular Infections: Multicenter Data From Turkey
Brief Title: Analysis of Candida-Associated Osteoarticular Infections: Multicenter Turkish Data
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Collaborators: Istinye University (Other)
Responsible Party: Principal Investigator, Özlem Güler, Assistant Professor M.D., Kocaeli University
Other Study IDs: GOKAEK-2024/04.05 2024/40
Record Dates: First submitted 2024-12-04; First posted 2025-01-23 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Candida Osteomyelitis; Candida Infection; Arthritis; Spondylodiskitis
MeSH Terms: conditions — Candidiasis; Arthritis; Discitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Candida osteoarticular infections: Patients with an osteoarticular infection diagnosed on the basis of Candida growth in deep tissue culture, bone or joint fluid, and clinical and radiologic findings.

SUMMARY:
The aim of this observational study was to retrospectively analyze the osteoarticular infections caused by Candida spp. in adult patients in Turkey during the last decade and to determine the distribution of causative agents, demographic data, risk factors, clinical, radiological and laboratory findings. It was also aimed to compare treated and untreated cases and to reveal the factors influencing the success of treatment.

DETAILED DESCRIPTION:
Osteoarticular infections caused by Candida species can cause serious morbidity if not diagnosed and treated early. There are two large reviews of osteomyelitis and arthritis cases in the literature, and other data on the disease are based on case reports or small case series. Treatment recommendations for rare infections, such as Candida-associated osteomyelitis, are based on small case series and case reports from randomized clinical trials designed on other clinical forms of the disease. Amphotericin B is the most commonly used treatment of choice; however, recent reports suggest that fluconazole or echinocandin may be used. There are case reports in Turkey, but no multicenter study data have been reported.

The aim of this retrospective observational study was to investigate the osteoarticular infections caused by Candida spp. in Turkey, to reveal the distribution of causative agents, demographic data, risk factors, clinical, radiologic and laboratory findings, and to contribute to the literature with the data to be obtained at the end of the study in the management of these infections by comparing successful and unsuccessful cases in treatment.

It was planned to share the Excel file prepared by the principal investigator containing the data to be collected via e-mail, and to evaluate all the data after collection via e-mail.

Statistical evaluation will be performed using IBM SPSS (version 29.0; IBM Corp., Armonk, NY, USA). Chi-square and Fisher's exact tests will be used to compare the categorical variables. The conformity of measurement variables to normal distribution will be examined by Kolmogorov-Smirnov test. Descriptive analyses will be presented using the mean, standard deviation, median, and minimum-maximum values. Risk factors for treatment failure or side effects will be evaluated using the Mann-Whitney U test or Student's t-test. Treatment failure will be considered the dependent variable and will be analyzed using univariate logistic regression with other variables. A P value < 0.05 will be considered significant. In a stepwise approach, the variables found to be significant in the univariate logistic regression test will be analyzed using multivariate logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age
2. Cases of osteomyelitis, septic arthritis and spondylodiscitis due to Candida spp.
3. Deep tissue culture, joint fluid or bone tissue growth is required. In addition, patients with compatible clinical and radiographic findings will be enrolled.

Exclusion Criteria:

1. Pediatric patients
2. Patients with Candida spp. growth in superficial tissue culture will not be part of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Since it is a rare disease, all cases reported from various centers in Turkey will be included. Efforts will be made to reach as many centers as possible through the mailing lists.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
The aim of this study was to evaluate the clinical findings of patients with Candida osteoarticular infection. | Data will be collected retrospectively by reviewing the files of cases diagnosed in the last ten years (between 1 January 2014 and 1 December 2024) (last 10 years). Review of files and enrollment of cases into the study started on 5 December 2024.
  Description This outcome measure aims to assess the findings of cases of Candida osteoarticular infection. Four specific findings will be inquired about.
  Pain, swelling, redness, and purulent discharge.
  Measurement Tool/Method: Clinical findings will be assessed using a patient chart review form.
  Unit of Measure: Each clinical finding will be expressed as a percentage.
Microbiological Characteristics of Candida species | Data will be collected retrospectively by reviewing the files of cases diagnosed in the last ten years (between 1 January 2014 and 1 December 2024) (last 10 years). Review of files and enrollment of cases into the study started on 5 December 2024.
  Description: This outcome measure aims to describe the microbiological profiles of Candida osteoarticular infections
  Measure Description Fungal culture results by VITEC-2 or MALDI-TOF will be evaluated.
  Unit of measurement: Percentage of Candida species detected.

SECONDARY OUTCOMES:
Treatment success of Candida osteoarticular infections | Data will be collected retrospectively by reviewing the files of cases diagnosed in the last ten years (between 1 January 2014 and 1 December 2024) (last 10 years). Review of files and enrollment of cases into the study started on 5 December 2024.
  This outcome measure investigates the success rate of treatment strategies for Candida osteoarticular infections. Treatment success is defined as resolution of symptoms, eradication of infection, and no recurrence within 6 months after completing therapy.
  Measurement Tool/Method: Success will be assessed based on follow-up clinical evaluations and microbiological clearance confirmed by repeat cultures.
  Unit of Measure: Percentage of participants achieving treatment success.

OTHER OUTCOMES:
Factors affecting treatment success | Data will be collected retrospectively by reviewing the files of cases diagnosed in the last ten years (between January 1, 2014, and December 1, 2024) (the last 10 years). The review of files and the enrollment of cases into the study by invitation began
  Factors affecting treatment success The evaluation will be conducted using the logistic regression method. The results will be presented as an odds ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Güler, Asst. Prof., Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with infectious disease physicians and academics for a period of two years following the release of the study protocol
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data can be shared for two years after study protocol release
Access Criteria: Infectious disease physicians access is appropriate

REFERENCES:
- [Background] Gamaletsou MN, Kontoyiannis DP, Sipsas NV, Moriyama B, Alexander E, Roilides E, Brause B, Walsh TJ. Candida osteomyelitis: analysis of 207 pediatric and adult cases (1970-2011). Clin Infect Dis. 2012 Nov 15;55(10):1338-51. doi: 10.1093/cid/cis660. Epub 2012 Aug 21. PMID 22911646
- [Background] Gamaletsou MN, Rammaert B, Bueno MA, Sipsas NV, Moriyama B, Kontoyiannis DP, Roilides E, Zeller V, Taj-Aldeen SJ, Miller AO, Petraitiene R, Lortholary O, Walsh TJ. Candida Arthritis: Analysis of 112 Pediatric and Adult Cases. Open Forum Infect Dis. 2015 Dec 23;3(1):ofv207. doi: 10.1093/ofid/ofv207. eCollection 2016 Jan. PMID 26858961
- [Background] Pappas PG, Kauffman CA, Andes DR, Clancy CJ, Marr KA, Ostrosky-Zeichner L, Reboli AC, Schuster MG, Vazquez JA, Walsh TJ, Zaoutis TE, Sobel JD. Clinical Practice Guideline for the Management of Candidiasis: 2016 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2016 Feb 15;62(4):e1-50. doi: 10.1093/cid/civ933. Epub 2015 Dec 16. PMID 26679628